CLINICAL TRIAL: NCT06712004
Title: Efficacy and Safety of Bevifibatide Citrate Injection in Patients With Acute Ischemic Stroke Without Large or Medium-Sized Vessel Occlusion: A Single-Center, Randomized, Double-Blind, Dose-Response Controlled Clinical Trial
Brief Title: A Dose-Response Controlled Trial of Bevifibatide for Acute Ischemic Stroke
Acronym: BCAIS-I
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LC2024ZD032
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke, Acute; Ischemic Stroke; Cerebral Infarction; Brain Diseases
Keywords: Bevifibatide citrate injection; Dose-response controlled; Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke; Cerebral Infarction; Brain Diseases

STUDY DESIGN:
Intervention Model Description: The subject numbers and corresponding medication numbers are permanently identified and unique for each successfully randomized patient. If any patients who have been successfully randomized do not receive the trial medication or cannot be reassigned to others, their medication and medication numbers will be invalidated by the medication administrator. To ensure blinding during the trial execution, unblinded personnel responsible for administering and configuring the trial drug must sign a confidentiality agreement. Investigators, other blinded investigators, subjects, and sponsors will not have access to any information regarding group assignment or related documents pertaining to the trial drug.
Who Masked: Participant, Investigator
Masking Description: The subject numbers and corresponding medication numbers are permanently identified and unique for each successfully randomized patient. If any patients who have been successfully randomized do not receive the trial medication or cannot be reassigned to others, their medication and medication numbers will be invalidated by the medication administrator. To ensure blinding during the trial execution, unblinded personnel responsible for administering and configuring the trial drug must sign a confidentiality agreement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine maintenance dose group (Experimental): Undergoing bevifibatide citrate injection with intravenous bolus of 220μg/kg (0.11ml/kg) over 1 to 2 minutes, followed by continuous intravenous bolus at a rate of 2.5μg/kg/min (0.075ml/kg/h) for 24 hours.
  Interventions: Drug: Bevifibatide citrate injection
- Low maintenance dose group (Experimental): Undergoing bevifibatide citrate injection with intravenous bolus of 220μg/kg (0.11ml/kg) over 1 to 2 minutes, followed by continuous intravenous bolus at a rate of 2.0μg/kg/min (0.06ml/kg/h) for 24 hours.
  Interventions: Drug: Bevifibatide citrate injection

INTERVENTIONS:
Drug: Bevifibatide citrate injection — Bevifibatide citrate injection should be diluted with 0.9% NaCl solution. After the completion of the study drug infusion, if a follow-up cranial NCCT/MRI within 48 hours shows no significant intracranial hemorrhage, all patients will be administered enteric-coated aspirin tablets (100mg, qd) and clopidogrel hydrogen sulfate tablets (75mg, qd) until day 90. All patients will be managed in accordance with the current guidelines for stroke management. The use of low molecular weight heparin for the prevention of deep vein thrombosis is permitted.
  Other Names: BETAGRIN

SUMMARY:
BCAIS-I is a single-center, randomized, double-blind, dose-response controlled clinical Trial, to preliminarily explore the efficacy of two different maintenance doses of bevifibatide citrate injection in improving 90-day neurological outcomes and the incidence of symptomatic intracranial hemorrhage in patients with acute ischemic stroke without large or medium-sized vessel occlusion, aiming to identify a dosing regimen that maintains therapeutic efficacy while minimizing the rates of symptomatic intracranial hemorrhage and serious adverse events, thereby providing dosing evidence for future large-scale randomized controlled trials.

DETAILED DESCRIPTION:
Bevifibatide is a derivative similar to Eptifibatide, differing by only one amino acid: in the position where Eptifibatide contains high arginine, it is replaced by arginine to form Bevifibatide. Bevifibatide can specifically bind to the GPIIb/IIIa receptor, inhibiting platelet aggregation or adhesion. It also inhibits the integrin receptor αvβ3, thereby suppressing the growth of vascular smooth muscle and playing an important role in preventing arterial re-occlusion. Bevifibatide is a post-marketing product indicated for unstable angina, non-Q wave myocardial infarction, non-ST segment elevation myocardial infarction, and anti-thrombotic therapy during and around percutaneous coronary intervention. Its clinical formulation is an injectable solution for intravenous administration. When Bevifibatide is used in combination with clinical baseline medications, it has a synergistic effect on anti-platelet aggregation. Early oral administration of aspirin and clopidogrel can achieve a rapid synergistic effect on anti-platelet aggregation.

Currently, there are no clinical trials assessing the relationship between the dosage of Bevifibatide and its efficacy in treating acute ischemic stroke. We conduct a single-center, randomized, double-blind, dose-response controlled clinical trial to preliminarily evaluate and compare the effectiveness of conventional dosage and low maintenance dosage of Bevifibatide citrate injection in improving neurological outcomes at 90 days and the incidence of symptomatic intracranial hemorrhage in patients suffering from acute ischemic stroke without large or medium-sized vessel occlusion, thereby determining a relatively safe dosage while maintaining the effectiveness of the medication, and providing a dosage basis for conducting large-sample randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Any of the following presentations of acute ischemic stroke (AIS): ① Within 24 hours of time last known well and ineligible for intravenous thrombolysis (IVT) or endovascular treatment (EVT). ② More than 24 hours and less than 96 hours after time last known well but within 24 hours of ischemic stroke progression [worsening of ≥ 2 points on the NIHSS]; and ineligible for IVT or EVT without ICH confirmed by CT scan or MRI. ③ Treated with IVT followed by early neurological deterioration (worse NIHSS by ≥ 4 points) within the first 24 hours after IVT without ICH confirmed by CT scan or MRI. ④ Treated with IVT followed by no neurological improvement (Neurological improvement is defined as decrease in the NIHSS score by ≥ 2 points) from baseline within 4 to 24 hours after IVT without ICH confirmed by CT scan or MRI.
* NIHSS score ≥ 3 immediately prior to trial entry.
* Without visible large or medium intracranial vessel occlusion on CT angiography (CTA), MR angiography (MRA), or digital subtraction angiography (DSA). (Qualifying mechanisms are: 1. hypoperfusion caused by arterial stenosis; 2. the initial occluded large or medium artery spontaneously recanalized or recanalized with IVT before the vascular imaging performed; 3. multiple or single distal emboli from cardiac or other sources in arterial branches too small to visualized on CTA or MRA; 4. lacunar infarct due to small vessel occlusion).
* Written informed consent obtained from patients or their legal representatives.

Exclusion Criteria:

* CT or MR evidence of intracranial haemorrhage.
* Pre-morbid disability with a mRS score ≥ 2.
* Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, sick sinus syndrome, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within three months, dilated cardiomyopathy, left atrial spontaneous echo contrast, ejection fraction less than 30%.
* Planned treatment with dual antiplatelet therapy within 1week of the index stroke.
* Any history of a primary or other intracerebral (parenchymal) haemorrhage (intraventricular, subarachnoid, subdural, epidural).
* Any untreated or incompletely treated intracranial aneurysm, any intracranial vascular malformation or any intracranial tumour.
* Currently pregnant or lactating, and those planned to conceive.
* Subjects with positive urine HCG test results.
* Known allergy to study medication or concomitant medications.
* Gastrointestinal bleeding, urinary tract bleeding, or other major systemic haemorrhage within 30 days.
* Any major surgery within 6 weeks of the index stroke.
* History of heparin-induced thrombocytopenia.
* Expected lifespan less than 3 months.
* Pre-existing neurological or psychiatric disease that would confound the neurological functional outcome evaluations.
* Any of the following laboratory tests: INR [International Normalized Ratio]>2.0, PT>1.3 times normal value, platelet count<100 × 109/L, Hb<10g/dl.
* Systolic pressure greater than 180 mmHg or diastolic pressure greater than 110 mmHg after aggressive treatment.
* Severe renal insufficiency (glomerular filtration rate < 30 ml/min or serum creatinine > 220 μmol/L [2.5 mg/dl]).
* History of liver dysfunction (AST/ALT exceeding the upper limit of normal by more than twice) or cirrhosis.
* Arterial tortuosity and/or other arterial diseases that prevent the expected internal thrombectomy device from reaching the target vessel.
* Unlikely to be available for 90-day follow-up.
* Current participation in another treatment clinical trial.
* Other conditions that are not suitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale (mRS) score | 90(±7) days
  The mRS scores are evaluated by experienced researchers trained in standard neurological function assessments using information obtained from patients or their families.
Symptomatic intracranial hemorrhage (sICH) | Within 48 hours
  ICH will be evaluated according to the Heidelberg Bleeding Classification. sICH is diagnosed if the new observed ICH is associated with any of the following conditions: 1) NIHSS score increased more than 4 points than that immediately before worsening; 2) NIHSS score increased more than 2 points in one category; 3) Deterioration led to intubation, hemicraniectomy, external ventricular drain placement or any other major interventions. Additionally, the symptom deteriorations could not be explained by causes other than the observed ICH.

SECONDARY OUTCOMES:
mRS score 0-1 at 30 days | 30(±3) days
  Proportion of patients without disability at 30 days.
mRS score 0-2 at 30 days | 30(±3) days
  Proportion of patients with functional independence at 30 days.
mRS score 0-1 at 90 days | 90(±7) days
  Proportion of patients without disability at 90 days.
mRS score 0-2 at 90 days | 90(±7) days
  Proportion of patients with functional independence at 90 days.
Change of the National Institute of Health Stroke Scale (NIHSS) score from baseline to 72 hours | 72(±12) hours
  Change of the NIHSS score from baseline to 72 hours
Change of the NIHSS score from baseline to 6 days | 6(±1) days
  Change of the NIHSS score from baseline to 6 days
Change of the NIHSS score from baseline to 90 days | 90(±7) days
  Change of the NIHSS score from baseline to 90 days
Health-related quality of life | 90(±7) days
  Health-related quality of life is assessed with the European Quality Five Dimensions Five Level scale (EQ-5D-5L)
Any ICH | Within 48 hours
  ICH will be evaluated according to the Heidelberg Bleeding Classification.
Mortality | 90(±7) days
  Mortality rates are defined as the number of deaths observed divided by the number of subjects observed over the 90-day study period.
Incidence of serious adverse events | 90(±7) days
  Including both bleeding and non-bleeding adverse events. Among these, bleeding adverse events encompass: purpura, minor oral and nasal mucosal bleeding, ecchymosis, gingival bleeding, epistaxis, minor gastrointestinal or urinary tract bleeding, hematomas from spontaneous or minor trauma, hemarthrosis, intracranial hemorrhage, and bleeding that poses hemodynamic compromise or requires intervention.
  Serious adverse events are defined as undesirable medical events that occur after a subject has received the investigational product, including death, life-threatening conditions, permanent or significant disability, or loss of function, hospitalization or prolongation of hospital stay due to the event, and congenital anomalies or birth defects.
Incidence of adverse events | 90(±7) days
  Including both bleeding and non-bleeding adverse events. Among these, bleeding adverse events encompass: purpura, minor oral and nasal mucosal bleeding, ecchymosis, gingival bleeding, epistaxis, minor gastrointestinal or urinary tract bleeding, hematomas from spontaneous or minor trauma, hemarthrosis, intracranial hemorrhage, and bleeding that poses hemodynamic compromise or requires intervention.
  Adverse events are defined as any harmful or unintended responses occurring in a clinical trial that may be related to the investigational product. There should be at least a reasonable possibility of a causal relationship between the study product and the adverse reaction, meaning that a connection cannot be ruled out.
Inhibitory rate of platelet aggregation at 4 hours | 4 hours
  ADP-induced platelet aggregation.
Inhibitory rate of platelet aggregation at 24 hours | 24 hours
  ADP-induced platelet aggregation.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanzhi Duan, MD, Study Director — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No